CLINICAL TRIAL: NCT01248871
Title: "Volatile Anesthetic Protection Of Renal Transplants: VAPOR-1-trail
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VAPOR 001
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Kidney Donation/Transplantation
Keywords: renal; transplantation; Volatile; anesthetic
MeSH Terms: interventions — Sufentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- SEVO (Active Comparator): sevoflurane-remifentanil/sufentanil combination
  Interventions: Drug: procedure:sevoflurane-remifentanil/sufentanil
- SERE (Active Comparator): volatile agent only during reperfusion
  Interventions: Drug: volatile agent only during reperfusion
- propofol (Active Comparator): propofol-remifentanil/sufentanil
  Interventions: Drug: propofol-remifentanil/sufentanil

INTERVENTIONS:
Drug: procedure:sevoflurane-remifentanil/sufentanil — Active Comparator
  Arms: SEVO
Drug: volatile agent only during reperfusion — Active Comparator
  Arms: SERE
Drug: propofol-remifentanil/sufentanil — Active Comparator
  Arms: propofol

SUMMARY:
To compare the renal protective properties of two currently used anaesthetic techniques - a sevoflurane-remifentanil/sufentanil combination with a propofol-remifentanil/sufentanil combination for anaesthesia in patients undergoing living donor kidney donation/transplantation.

ELIGIBILITY:
Inclusion Criteria:

* All patients: Age > 18 years

Exclusion Criteria:

* patient refusal
* BMI< 17, >35
* neurological disorder
* recent use of psycho-active medication, including alcohol.
* Donor-recipient couples from the ABO-incompatible program
* Altruistic donor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To compare the renal protective properties of two currently used anaesthetic techniques | participants will be followed for the duration of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: M.M.R.F Struys, Prof.dr., Principal Investigator — University Medical Center Groningen; R,J. Ploeg, Prof.dr, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Nieuwenhuijs-Moeke GJ, Nieuwenhuijs VB, Seelen MAJ, Berger SP, van den Heuvel MC, Burgerhof JGM, Ottens PJ, Ploeg RJ, Leuvenink HGD, Struys MMRF. Propofol-based anaesthesia versus sevoflurane-based anaesthesia for living donor kidney transplantation: results of the VAPOR-1 randomized controlled trial. Br J Anaesth. 2017 May 1;118(5):720-732. doi: 10.1093/bja/aex057. PMID 28510740